CLINICAL TRIAL: NCT01875991
Title: An Open-label, Randomized, Crossover Study to Assess the Preference for Autoinjector A Versus Autoinjector B in Rheumatoid Arthritis and Plaque Psoriasis Subjects Treated With Etanercept
Brief Title: Preference Between Two Autoinjectors in Patients With Rheumatoid Arthritis and Plaque Psoriasis Treated With Etanercept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20090176
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis; Plaque Psoriasis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autoinjector A (Experimental): Participants self-injected 50 mg etanercept once a week (RA) or twice a week (PsO) using Autoinjector A for 4 weeks.
  Interventions: Drug: Etanercept via Autoinjector A
- Autoinjector B (Experimental): Participants self-injected 50 mg etanercept once a week (RA) or twice a week (PsO) using Autoinjector B for 4 weeks.
  Interventions: Drug: Etanercept via Autoinjector B

INTERVENTIONS:
Drug: Etanercept via Autoinjector A — Autoinjector A is a hand-held, reusable, electromechanical device used with a single-use disposable cassette preassembled with an etanercept 50-mg prefilled syringe.
  Arms: Autoinjector A
Drug: Etanercept via Autoinjector B — Autoinjector B is a single-use, spring-loaded, self-contained autoinjector preassembled with an etanercept 50-mg prefilled syringe.
  Other Names: Enbrel® SureClick®
  Arms: Autoinjector B

SUMMARY:
The study will estimate the preference of rheumatoid arthritis (RA) and Plaque Psoriasis (PsO) patients who self inject etanercept for one of two experimental autoinjectors.

DETAILED DESCRIPTION:
Candidates for treatment are those who in the determination of the investigator's standard of care and the caring physician's intent are to initiate treatment with etanercept. Participants must be naïve to etanercept and naïve to other autoinjector pens or prefilled syringes and be able to self-inject. The study will consist of a 30 day screening period, and 2 treatment periods of 4 weeks duration each (one treatment period using Autoinjector A and the other using Autoinjector B). At the end of the study, participants may continue treatment with commercially available etanercept at the physician's discretion.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of moderate to severe Rheumatoid Arthritis (RA) or moderate to severe Plaque Psoriasis (PsO) and a candidate for treatment with etanercept in the opinion of the investigator in addition to the caring physician's intent to initiate treatment with etanercept. - Naive to etanercept. - Naive to other autoinjector pens or prefilled syringes for Tumor Necrosis Factor (TNF)-inhibitor therapy or other subcutaneous biologics for RA. - Willing to self-inject per investigator judgement at screening and capable of self-injection using the autoinjector A or B as documented at baseline by the investigator. - Able to read and write in English. -

Exclusion Criteria: Latex allergy. - Subject has an active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to first dose of etanercept. - Subject had prosthetic joint infection within 5 years of screening or native joint infection within 1 year of screening.

* Other criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2013-06-05 (Actual); Primary Completion 2014-03-04 (Actual); Study Completion 2014-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (37):
- United States (28):
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, San Diego, California
  - Research Site, San Ramon, California
  - Research Site, Santa Maria, California
  - Research Site, Tustin, California
  - Research Site, Denver, Colorado
  - Research Site, Dunedin, Florida
  - Research Site, Tampa, Florida
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Lansing, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Orchard Park, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Hixson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Clarksburg, West Virginia
- Canada (9):
  - Research Site, Victoria, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Barrie, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Peterborough, Ontario

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults (≥ 18 years) with moderate to severe rheumatoid arthritis (RA) or plaque psoriasis (PsO) and candidates for treatment with etanercept (Enbrel) in the opinion of the investigator in addition to the caring physician's intent to initiate treatment with etanercept.
  First patient enrolled on 05 June 2013; last patient enrolled 03 January 2014.
Pre-assignment Details: Randomization was stratified by disease state (RA and PsO). Each participant served as his or her own control in this crossover study.
Groups:
- Autoinjector A / Autoinjector B: Participants self-injected 50 mg etanercept once a week (RA) or twice a week (PsO) using Autoinjector A for 4 weeks, and then switched over to Autoinjector B for an additional 4 weeks of treatment.
- Autoinjector B / Autoinjector A: Participants self-injected 50 mg etanercept once a week (RA) or twice a week (PsO) using Autoinjector B for 4 weeks, and then switched over to Autoinjector A for an additional 4 weeks of treatment.
Period: Overall Study
Arm/Group | Autoinjector A / Autoinjector B | Autoinjector B / Autoinjector A
Started | 108 | 109
Received Etanercept in Period 1 | 108 | 108
Received Etanercept in Period 2 | 102 | 103
Completed | 101 | 103
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autoinjector A / Autoinjector B | Autoinjector B / Autoinjector A | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (13.8) | 53.2 (13.6) | 54.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 34 | 35 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Black or African American | 5 | 3 | 8
  White | 100 | 102 | 202
  Other | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 99 | 99 | 198
Disease State [Number; unit: participants]
  Rheumatoid Arthritis | 79 | 78 | 157
  Plaque Psoriasis | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Preference for Autoinjector A Versus Autoinjector B
Description: Preference for autoinjector A versus autoinjector B was assessed by Question 1 of the Subject Preference Questionnaire administered after the completion of the 2 treatment periods at Week 8. Participants answered the question "Which autoinjector do you prefer overall?"
Time Frame: Week 8
Population: The primary analysis set consisted of all randomized participants who received at least 1 injection of Eetanercept with each autoinjector and indicated a preference for an autoinjector in the Subject Preference Questionnaire. N = number of participants with RA and PsO respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Primary Analysis Set: Participants who received at least one injection with each autoinjector and completed the Subject Preference Questionnaire.
Arm/Group | Primary Analysis Set
Number analyzed (Participants) | 204
percentage of participants
  Overall | 41.7 [34.9 to 48.4]
  Rheumatoid Arthritis (N=147) | 43.5 [35.5 to 51.6]
  Plaque Psoriasis (N=57) | 36.8 [24.3 to 49.4]

2. Secondary Outcome: Change From Baseline in Needle Apprehension at Week 4
Description: Participants' needle apprehension was assessed using the Subject's Perception of Self-Injecting Questionnaire. Participants answered the question "Overall how nervous are you about the needle when you think about giving yourself etanercept using the autoinjector" using a scale from 1 (extremely nervous) to 5 (not at all nervous).
Time Frame: Baseline and Week 4
Population: Full analysis set, which included all randomized participants. "n" indicates the number of participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 108 | 109
units on a scale
  Baseline (n=108, 109) | 3.94 (0.96) | 4.00 (1.02)
  Change from Baseline (n= 102, 106) | 0.31 (1.01) | 0.39 (0.91)
Statistical Analysis 1: Comparison: Autoinjector A vs Autoinjector B; Test type: Superiority or Other; p = 0.501, Van Elteren test; P-value for 'All subjects' from Van Elteren test adjusting for strata (RA or PsO)

3. Secondary Outcome: Ease of Use
Description: Ease of use was assessed based on responses to questions 1 to 6 of the Subject's Experience with the Autoinjector Questionnaire: 1. How easy was it to learn how to use the autoinjector? 2. How easy was it for you to press the button to start the injection? 3. How easy was the autoinjector to use? 4. How easy was it to hold the autoinjector throughout the injection? 5. How easy was it for you to inject yourself using the autoinjector? 6. How easy was it to follow the progress of the injection? Each question was answered on a scale from 1 (Very difficult) to 5 (Very easy). The percentage of participants who scored either a 4 (Somewhat easy) or 5 (Very easy) on each question is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 207
percentage of participants
  Ease of learning how to use the autoinjector | 92.3 | 96.1
  Ease of pressing button to start the autoinjector | 95.7 | 90.8
  Ease of using the autoinjector | 91.3 | 88.9
  Ease of holding the autoinjector | 89.4 | 88.4
  Ease of self-injecting | 88.0 | 87.0
  Ease of following progress | 94.2 | 87.4

4. Secondary Outcome: Certainty of Completing the Injection With the Autoinjector
Description: Certainty of completing the injection with the autoinjector was assessed based on responses to Question 7 of the Subject's Experience with the Autoinjector Questionnaire: "How certain were you that you knew when the injection was finished?" Participants answered on a scale from 1 (Not at all) to 5 (Extremely). The percentage of participants who scored 4 (Very) or 5 (Extremely) is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 206
percentage of participants | 94.2 | 87.9

5. Secondary Outcome: Convenience
Description: Convenience was assessed based on responses to Question 8 of the Subject's Experience with the Autoinjector Questionnaire: "How convenient was the autoinjector to use?" Participants answered on a scale from 1 (Not at all) to 5 (Very much). The percentage of participants who scored a 4 (Quite a bit) or 5 (Very much) is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 207
percentage of participants | 76.9 | 86.5

6. Secondary Outcome: Discomfort
Description: Discomfort was assessed based on responses to Question 9 of the Subject's Experience with the Autoinjector Questionnaire: "How much discomfort did you experience when giving yourself the medicine using the autoinjector?" Participants answered on a scale from 1 (None) to 5 (Very much). The percentage of participants who scored a 1 (None) or 2 (A little) is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 207
percentage of participants | 56.3 | 72.5

7. Secondary Outcome: Satisfaction
Description: Satisfaction was assessed based on responses to questions 11 and 12 of the Subject's Experience with the Autoinjector Questionnaire. Question 11: "How dependable (durable, sturdy, reliable) did you feel the autoinjector device was?" answered on a scale from 1 (Not at all) to 5 (Very much). Question 12: "Overall, how likely would you be to recommend the autoinjector to someone like you who is on etanercept?" answered on a scale from 1 (Would not recommend) to 5 (Highly likely to recommend). The percentage of participants who scored either a 4 or 5 on each question is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 207
percentage of participants
  How dependable did you feel | 79.8 | 86.0
  Likeliness of recommending autoinjector | 66.8 | 84.5

8. Secondary Outcome: Pain Associated With Use of the Autoinjector
Description: Pain associated with use of the autoinjector was assessed based on responses to Question 10 of the Subject's Experience with the Autoinjector Questionnaire: "Using this scale, select the circle that best describes how much it hurt when giving yourself an injection." Participants answered on a scale from 0 (No hurt) to 5 (Hurts worst). The percentage of participants who scored a 0 (No hurt) or 1 (Hurts a little bit) is reported.
Time Frame: At the end of each treatment period; Week 4 and Week 8
Population: Full analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Autoinjector A | Autoinjector B
Number analyzed (Participants) | 208 | 207
percentage of participants | 51.4 | 65.2

9. Secondary Outcome: Strength of Preference for Autoinjector A and Autoinjector B
Description: Strength of preference for Autoinjector A versus Autoinjector B was assessed by Question 2 of the Subject Preference Questionnaire administered after the completion of the two treatment periods at Week 8. After selecting which autoinjector they preferred overall, participants were asked to indicate how much they preferred it on a scale from 1 (Slightly), 2 (Somewhat), 3 (Strongly) and 4 (Vey Strongly).
Time Frame: Week 8
Population: Primary Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- Autoinjector A Preference: Participants who preferred Autoinjector A overall
- Autoinjector B Preference: Participants who preferred Autoinjector B overall
Arm/Group | Autoinjector A Preference | Autoinjector B Preference
Number analyzed (Participants) | 85 | 119
percentage of participants
  Very Strongly | 45.9 [34.9 to 48.4] | 36.1
  Strongly | 43.5 [35.5 to 51.6] | 41.2
  Somewhat | 5.9 [24.3 to 49.4] | 16.8
  Slightly | 4.7 | 5.9

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Autoinjector A | Autoinjector B
Serious Adverse Events (participants affected / at risk) | 9/211 | 2/210
Other Adverse Events (participants affected / at risk) | 12/211 | 6/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autoinjector A (N=211) | Autoinjector B (N=210)
Atrial flutter (Cardiac disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autoinjector A (N=211) | Autoinjector B (N=210)
Injection site erythema (General disorders) | 12 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.